CLINICAL TRIAL: NCT02925260
Title: Pelvic Collections on MRI in Patients With Ileal Pouches, and a Feasibility Study of Dynamic MRI Enema and Defaecating MRI Pouchography
Brief Title: MRI in Normal Ileal Pouches, and a Feasibility Study of Dynamic MRI Enema and Defaecating MRI Pouchography
Status: Completed | Type: Observational
Sponsor: London North West Healthcare NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: mripouchesv1.11808216
Record Dates: First submitted 2016-10-03; First posted 2016-10-05 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Colitis, Ulcerative; Ileal Pouches
MeSH Terms: conditions — Colitis, Ulcerative | interventions — Magnetic Resonance Spectroscopy; Enema

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with normal ileal pouches: Inclusion Criteria
  * Ileal pouch reservoir in situ
  * Greater than three years since closure of ileostomy
  * Normal pouch function as defined by Orësland score of <4
  * Never had a diagnosis of pouchitis
  * Never had treatment for pouchitis
  * No evidence of pouchitis on rigid pouchoscopy
  * CRP <10
  Interventions: Other: MRI with ileal pouch contrast and enema.

INTERVENTIONS:
Other: MRI with ileal pouch contrast and enema. — Pre enema 20mg IV or IM Hyoscine Butylbromide (Buscopan) Pre enema Small Field of View (SFOV) T2 sagittal series Pre enema SFOV T2 axial series Pre enema SFOV T1 sagittal series (fat suppressed) Pre enema SFOV T1 axial series (fat suppressed) Enema infiltration started During enema filling Dynamic T1 sagittal single image, fat suppressed, aligned on pouch-anal anastomosis During enema filling T1 sagittal series (fat suppressed) During enema filling T1 axial series (fat suppressed) Jelly infiltrated and held Evacuating series Oblique sagittal T2 evacuating series of the mid and distal pouch, aligned to the pouch-anal anastomosis

SUMMARY:
A study to investigate the prevalence of pelvic collections in a representative sample of participants with normally functioning ileal pouches. It also aims to establish the feasibility and reporting variables for dynamic MRI enemas in ileal pouches and defaecating enema pouchography.

DETAILED DESCRIPTION:
Ulcerative Colitis Ulcerative Colitis (UC) is the most common of the inflammatory bowel diseases, with approximately 146,000 sufferers in the UK (NICE, 2011). Unlike other inflammatory bowel diseases, the inflammation in UC affects only the large bowel, starting at the rectum and extending proximally (towards the mouth end of the gut). Three in four patients are managed with medical treatments with acceptable control of their disease, but patients may require surgical removal of their large bowel for several reasons. The one in four patients who have their colon removed (colectomy) either need an emergency operation for infection, perforation or bleeding, or a planned operation for failure of medical management, intolerance to medication, cancer or steroid dependence (1). Because the inflammation is confined only to the colon, this surgery is curative.

Having removed the large bowel, there are options with regard to what to do with the end of the remaining small bowel, the ileum. In 1978 Professor Sir Alan Parks and Professor John Nicholls publicised their operation for 'restorative proctocolectomy' (RPC) folding and suturing together loops of small bowel to create a 'pouch' to take over the reservoir function of the rectum, and giving the patient the chance of continence without the need for a stoma (2,3). This operation has become extremely popular over the last 38 years, and is considered internationally to be the gold standard for 'restorative proctocolectomy' in patients who choose not to have a permanent stoma (4).

The operation has been refined in the years since it's introduction (5), with roughly two thirds of patients enjoying acceptable function. However, the complications associated with creating an RPC; notably pelvic sepsis, fistulae, poor mechanical function and inflammation, mean that the cumulative rate of pouch failure is roughly 5% at five years, and up to 15% at 15 years (Ryoo et al. 2014; Remzi et al. 2015; Sherman et al. 2014; R. et al. 2012; Papadopoulos et al. 2010).

Pouch-Related Septic Complications St Mark's Hospital has one of the largest UK cohorts of patients with RPCs, and is a tertiary referral centre for pouch complications. Of the reasons for pouch failure, chronic pelvic sepsis is the major cause, at 50 to 60%. This is a long term infection in the pelvis around or near the pouch, causing inflammation and poor function.

The pouch itself may become inflamed, known as pouchitis, and the cause for this is unknown, but it is hypothesised that the inflammation is caused by a change in the type of bacteria present in the pouch as opposed to the small bowel when it was in normal continuity.

Generally speaking, the management of pelvic sepsis causing pouch function is to surgically or radiologically drain the pelvic collection, or eventually surgically remove the pouch. The management of pouchitis (primary idiopathic pouchitis) is primarily with antibiotics, but in prolonged cases where antibiotics have been ineffective it may be in the patient's benefit to treat the inflammation with steroids or 'biologic' medications. These medications act by suppressing the body's innate immune response, and it would be inappropriate to use these medications if the true cause of inflammation is ongoing sepsis in the pelvis because this infection would likely become significantly worse, causing systemic infection (sepsis).

Unpublished research from St Mark's completed at the end of 2015 http://scripties.umcg.eldoc.ub.rug.nl/root/geneeskunde/2016/PloegVvander/ showed that in 68 patients treated for primary idiopathic pouchitis, 38% had an incidental pre-sacral collection identified on MRI, potentially consistent with pelvic sepsis driving the inflammation, rather than the inflammation rising primarily from the pouch itself.

Five patients went on to have drainage of the pelvic sepsis, with resolution of symptoms in only one. Therefore, based on this series, the significance of a pre-sacral collection on MRI in the context of pouchitis is unknown. Beyond this, it is not known how often this finding may be present as a 'normal variant' in patients with normal functioning pouches. The proposed trial would help to guide clinical management of patients with pouchitis and pre-sacral collections.

Pouch Evacuatory Dysfunction

A different type of problem with ileal pouches is the inability to easily evacuate the pouch. The majority of patients with normally functioning pouches, pressure to open their bowels is felt just like people with normal anatomy. Some patients have difficulty evacuating the pouch, often without an obvious inflammatory or anatomical cause. These patients are often investigated with defaecating pouchography, which is an investigation using moving x-ray images of radio-opaque contrast material being evacuated by the patient. A study conducted at St Mark's and published in August 2016 (11) demonstrated that this investigation has a relatively poor diagnostic value, partly due to the fact that there is no established range of normal findings. Using moving MRI images in patients with normal anatomy (called MRI defaecating proctography) is replacing the use of x-ray moving images (fluoroscopy) as there is as much, if not greater detail on the images, and there is no radiation exposure for the patient.

This study would be a pilot trial of the use of defaecating MRI in patients with pouches, (defaecating MRI pouchography) to establish whether the technique translates to patients with pouches instead of a rectum, and to establish what the range of normal findings are before going on to utilise the technique in patients with evacuatory dysfunction. This technique has not yet been described in the medical literature.

ELIGIBILITY:
Inclusion Criteria:

* • Ileal pouch reservoir in situ

  * Greater than three years since closure of ileostomy
  * Normal pouch function as defined by Orësland score of <4
  * Never had a diagnosis of pouchitis
  * Never had treatment for pouchitis
  * No evidence of pouchitis on rigid pouchoscopy
  * CRP <10

Exclusion Criteria:

* • Contraindications to magnetic resonance imaging (MRI) See appendix 1.

  * Unable or unwilling to agree to informed consent
  * Known inability to tolerate MRI (e.g. impaired mobility or claustrophobia)
  * Known gadolinium allergy
  * Known inability to maintain anal continence

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ulcerative colitis who have had an ileal pouch formed and never had any septic or inflammatory complications, at least three years from reversal of ileostomy.
Sampling Method: Non-Probability Sample
Enrollment: 19 (Actual)
Dates: Start 2017-05-10 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

PRIMARY OUTCOMES:
The prevalence of pelvic collections in a representative sample of patients with normally functioning ileal pouches. | Baseline ( MRI scan)

SECONDARY OUTCOMES:
A descriptive assessment of the normal variation of ileal pouches on MRI scans. | Baseline ( MRI scan)
Assess the patient experience of MRI pouchography using enemas | Baseline ( MRI scan)
  Non-validated questionnaire assessment of patient anxiety, comfort, embarrassment and confidence in the outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Guy HT Worley, BMBS MRCS, Principal Investigator — St. Mark's Hospital; Susan K Clark, PhD, Study Chair — St. Mark's Hospital
Locations (1):
- St Mark's Hospital, London, Middlesex, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Any data published will be fully anonymised. Identifiable patient data will be shared between the two sites conducting the research, this will be via secure email server. This arrangement is subject to UK Research and Ethics Committee scrutiny.

REFERENCES:
- [Background] Myrelid P, Oresland T. A reappraisal of the ileo-rectal anastomosis in ulcerative colitis. J Crohns Colitis. 2015 Jun;9(6):433-8. doi: 10.1093/ecco-jcc/jjv060. Epub 2015 Apr 11. PMID 25863275
- [Background] Oresland T, Bemelman WA, Sampietro GM, Spinelli A, Windsor A, Ferrante M, Marteau P, Zmora O, Kotze PG, Espin-Basany E, Tiret E, Sica G, Panis Y, Faerden AE, Biancone L, Angriman I, Serclova Z, de Buck van Overstraeten A, Gionchetti P, Stassen L, Warusavitarne J, Adamina M, Dignass A, Eliakim R, Magro F, D'Hoore A; European Crohn's and Colitis Organisation (ECCO). European evidence based consensus on surgery for ulcerative colitis. J Crohns Colitis. 2015 Jan;9(1):4-25. doi: 10.1016/j.crohns.2014.08.012. No abstract available. PMID 25304060
- [Background] NICE Centre for Clinical Practice. Ulcerative colitis: the management of ulcerative colitis. 2011;(June):1-68.
- [Background] Parks AG, Nicholls RJ. Proctocolectomy without ileostomy for ulcerative colitis. Br Med J. 1978 Jul 8;2(6130):85-8. doi: 10.1136/bmj.2.6130.85. PMID 667572
- [Background] Parks AG, Nicholls RJ, Belliveau P. Proctocolectomy with ileal reservoir and anal anastomosis. Br J Surg. 1980 Aug;67(8):533-8. doi: 10.1002/bjs.1800670802. PMID 7427044
- [Background] McLaughlin SD, Clark SK, Tekkis PP, Ciclitira PJ, Nicholls RJ. Review article: restorative proctocolectomy, indications, management of complications and follow-up--a guide for gastroenterologists. Aliment Pharmacol Ther. 2008 May;27(10):895-909. doi: 10.1111/j.1365-2036.2008.03643.x. Epub 2008 Feb 9. PMID 18266993
- [Background] Bach SP, Mortensen NJ. Revolution and evolution: 30 years of ileoanal pouch surgery. Inflamm Bowel Dis. 2006 Feb;12(2):131-45. doi: 10.1097/01.MIB.0000197547.80558.59. PMID 16432378
- [Background] Ryoo SB, Oh HK, Han EC, Ha HK, Moon SH, Choe EK, Park KJ. Complications after ileal pouch-anal anastomosis in Korean patients with ulcerative colitis. World J Gastroenterol. 2014 Jun 21;20(23):7488-96. doi: 10.3748/wjg.v20.i23.7488. PMID 24966620
- [Background] Remzi FH, Aytac E, Ashburn J, Gu J, Hull TL, Dietz DW, Stocchi L, Church JM, Shen B. Transabdominal Redo Ileal Pouch Surgery for Failed Restorative Proctocolectomy: Lessons Learned Over 500 Patients. Ann Surg. 2015 Oct;262(4):675-82. doi: 10.1097/SLA.0000000000001386. PMID 26366548
- [Background] Sherman J, Greenstein AJ, Greenstein AJ. Ileal j pouch complications and surgical solutions: a review. Inflamm Bowel Dis. 2014 Sep;20(9):1678-85. doi: 10.1097/MIB.0000000000000086. PMID 24983986
- [Background] Mennigen R, Senninger N, Bruewer M, Rijcken E. Pouch function and quality of life after successful management of pouch-related septic complications in patients with ulcerative colitis. Langenbecks Arch Surg. 2012 Jan;397(1):37-44. doi: 10.1007/s00423-011-0802-y. Epub 2011 May 19. PMID 21594657
- [Background] Papadopoulos VN, Michalopoulos A, Apostolidis S. Ileal pouch dysfunction. Tech Coloproctol. 2010 Nov;14 Suppl 1:S83-5. doi: 10.1007/s10151-010-0630-z. PMID 20725759
- [Background] Lovegrove RE, Tilney HS, Remzi FH, Nicholls RJ, Fazio VW, Tekkis PP. To divert or not to divert: A retrospective analysis of variables that influence ileostomy omission in ileal pouch surgery. Arch Surg. 2011 Jan;146(1):82-8. doi: 10.1001/archsurg.2010.304. PMID 21242450
- [Background] Sugerman HJ, Sugerman EL, Meador JG, Newsome HH Jr, Kellum JM Jr, DeMaria EJ. Ileal pouch anal anastomosis without ileal diversion. Ann Surg. 2000 Oct;232(4):530-41. doi: 10.1097/00000658-200010000-00008. PMID 10998651
- [Background] da Silva GM, Wexner SD, Gurland B, Gervaz P, Moon SD, Efron J, Nogueras JJ, Weiss EG, Vernava AM, Zmora O. Is routine pouchogram prior to ileostomy closure in colonic J-pouch really necessary? Colorectal Dis. 2004 Mar;6(2):117-20. doi: 10.1111/j.1463-1318.2004.00586.x. PMID 15008910
- [Background] Broder JC, Tkacz JN, Anderson SW, Soto JA, Gupta A. Ileal pouch-anal anastomosis surgery: imaging and intervention for post-operative complications. Radiographics. 2010 Jan;30(1):221-33. doi: 10.1148/rg.301095084. PMID 20083595
- [Background] Stellingwerf ME, Maeda Y, Patel U, Vaizey CJ, Warusavitarne J, Bemelman WA, Clark SK. The role of the defaecating pouchogram in the assessment of evacuation difficulty after restorative proctocolectomy and pouch-anal anastomosis. Colorectal Dis. 2016 Aug;18(8):O292-300. doi: 10.1111/codi.13431. PMID 27338231
- [Background] Flusberg M, Sahni VA, Erturk SM, Mortele KJ. Dynamic MR defecography: assessment of the usefulness of the defecation phase. AJR Am J Roentgenol. 2011 Apr;196(4):W394-9. doi: 10.2214/AJR.10.4445. PMID 21427302
- [Background] Nadgir RN, Soto JA, Dendrinos K, Lucey BC, Becker JM, Farraye FA. MRI of complicated pouchitis. AJR Am J Roentgenol. 2006 Oct;187(4):W386-91. doi: 10.2214/AJR.05.1019. PMID 16985109